CLINICAL TRIAL: NCT00285727
Title: Ropinirole Controlled Release (CR) as an Adjunctive Agent in the Treatment of Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Duke University (Other); GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2969
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Drug: Ropinirole CR

SUMMARY:
This is an 8 week study for patients who are currently taking antidepressant medication but not fully responding. Ropinirole CR would be taken in conjunction with current antidepressant medication. Patients come into the clinic once a week when starting on the medication and then once every other week for the remainder of the 8 weeks.

DETAILED DESCRIPTION:
We hope to learn whether ropinirole CR (controlled release formulation) is safe and effective when taken with an antidepressant to reduce the symptoms of depression. Adults who have a diagnosis of major depression and are currently taking an adequate dose of antidepressant medication will be sought for participation. They will continue to take the antidepressant medication and will receive ropinirole CR, an investigational medication, for eight weeks during which information will be collected about mood and cognitive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old
* Currently experiencing major depression
* On at least an adequate dose of fluoxetine, paroxetine, sertraline, citalopram, escitalopram, venlafaxine, bupropion, mirtazapine or duloxetine for at least 6 weeks (monotherapy). Exclusion Criteria:1. Pregnant females or females of child bearing years not using adequate birth control in the opinion of the investigators
* Known sensitivity to ropinirole
* Significant medical conditions that would preclude safe participation in the study in the opinion of the investigators.
* Significant abnormalities observed in screening laboratory evaluation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-01; Study Completion 2007-10

PRIMARY OUTCOMES:
HamD

SECONDARY OUTCOMES:
MADRS

CONTACTS AND LOCATIONS:
Overall Officials: Charles Debattista, Principal Investigator — Depression Research Clinic, Psychiatry Department, Stanford School of Medicine
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Depression Research Clinic, Psychiatry Department, Stanford School of Medicine, Stanford, California